CLINICAL TRIAL: NCT02615145
Title: Real World Evidence of the Effectiveness of Paritaprevir/r - Ombitasvir, ± Dasabuvir, ± Ribavirin in Patients With Chronic Hepatitis C - An Observational Study in Germany (LIFE-C)
Acronym: LIFE-C
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-398
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Results first posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic Hepatitis C; Dasabuvir; Ombitasvir+Paritaprevir+Ritonavir; Observational Study; Quality of life; Work-ability; Fibrosis; Cirrhosis
MeSH Terms: conditions — Hepatitis C, Chronic; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Genotype 1a (G1a) Participants: Treatment-naïve or -experienced participants with confirmed chronic hepatitis C (CHC) genotype 1a (G1a, includes all GT1-participants except participants with GT1b or GT1b/4), receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir with dasabuvir (ABBVIE REGIMEN) + ribavirin (RBV) according to standard of care and in line with the current local label.
  The prescription of a treatment regimen is at the discretion of the physician in accordance with local clinical practice and label, is made independently from this observational study and precedes the decision to offer the patient the opportunity to participate in this study.
- Genotype 1b (G1b) Participants: Treatment-naïve or -experienced participants with confirmed CHC genotype 1b (G1b; includes G1b/Genotype 4 [G4]), receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir with dasabuvir (ABBVIE REGIMEN) according to standard of care and in line with the current local label.
  The prescription of a treatment regimen is at the discretion of the physician in accordance with local clinical practice and label, is made independently from this observational study and precedes the decision to offer the patient the opportunity to participate in this study.
- Genotype 4 (G4) Participants: Treatment-naïve or -experienced participants with confirmed CHC genotype 4 (G4; non-G1), receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir (ABBVIE REGIMEN) + RBV according to standard of care and in line with the current local label.
  The prescription of a treatment regimen is at the discretion of the physician in accordance with local clinical practice and label, is made independently from this observational study and precedes the decision to offer the patient the opportunity to participate in this study.

SUMMARY:
The interferon-free combination regimen of paritaprevir/r - ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin (RBV) for the treatment of chronic hepatitis C (CHC) has been shown to be safe and effective in randomized controlled clinical trials with strict inclusion and exclusion criteria under well controlled conditions.

This observational study is the first effectiveness research examining the ABBVIE REGIMEN ± RBV, used according to local label, under real world conditions in Germany in a clinical practice patient population.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve or -experienced patients with confirmed CHC, genotype 1 or 4, receiving combination therapy with the interferon-free ABBVIE REGIMEN ± RBV according to standard of care and in line with local label.
* If RBV is co-administered with the ABBVIE REGIMEN, it has been prescribed in line with the current local label (with special attention to contraception requirements and contraindication during pregnancy)
* Patients must voluntarily sign and date a patient authorization to use and/or disclose his/her pseudonymized health data prior to inclusion into the study
* Patient must not be participating or intending to participate in a concurrent interventional therapeutic trial

Exclusion Criteria:

• Adolescents; people not treated according to label

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic Hepatitis C (CHC)
Sampling Method: Non-Probability Sample
Enrollment: 472 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ferenci P, Bourgeois S, Buggisch P, Norris S, Curescu M, Larrey D, Marra F, Kleine H, Dorr P, Charafeddine M, Crown E, Bondin M, Back D, Flisiak R. Real-world safety and effectiveness of ombitasvir/paritaprevir/ritonavir +/- dasabuvir +/- ribavirin in hepatitis C virus genotype 1- and 4-infected patients with diverse comorbidities and comedications: A pooled analysis of post-marketing observational studies from 13 countries. J Viral Hepat. 2019 Jun;26(6):685-696. doi: 10.1111/jvh.13080. Epub 2019 Mar 5. PMID 30739368
- See also: Related Info — http://rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this prospective, multi-center observational study, adult patients chronic hepatitis C (CHC) virus receiving the interferon-free ABBVIE REGIMEN (paritaprevir/r - ombitasvir with or without dasabuvir) with or without ribavirin (RBV) were offered the opportunity to participate in this study during a routine clinical visit at participating sites.
Pre-assignment Details: Per protocol, the Enrolled Population is used to present Participant Flow. Enrolled Population analysis groups are defined according to the participant's HCV genotype/subtype, regardless of ABBVIE Regimen prescribed.
Groups:
- Genotype 1a Participants: Treatment-naïve or -experienced participants with confirmed chronic hepatitis C (CHC) genotype 1a (G1a, includes all GT1- participants except participants with GT1b or GT1b/4), receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir with dasabuvir (ABBVIE REGIMEN) + ribavirin (RBV) according to standard of care and in line with the current local label.
- Genotype 1b Participants: Treatment-naïve or -experienced participants with confirmed CHC genotype 1b (G1b; includes G1b/G4), receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir with dasabuvir (ABBVIE REGIMEN) according to standard of care and in line with the current local label.
- Genotype 4 Participants: Treatment-naïve or -experienced participants with confirmed CHC genotype 4 (G4; non-G1), receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir (ABBVIE REGIMEN) + RBV according to standard of care and in line with the current local label.
- Missing: Treatment-naïve or -experienced participants with confirmed CHC but no genotype information.
Period: Overall Study
Arm/Group | Genotype 1a Participants | Genotype 1b Participants | Genotype 4 Participants | Missing
Started | 145 | 278 | 48 | 1
2 DAA + Ribavirin (RBV) (2 direct-acting antivirals (2DAA): paritaprevir/ritonavir - ombitasvir (ABBVIE REGIMEN) plus RBV) | 0 | 0 | 45 | 0
3DAA (3 direct-acting antivirals (3DAA): paritaprevir/ritonavir - ombitasvir + dasabuvir (ABBVIE REGIMEN)) | 5 | 261 | 0 | 0
3DAA + RBV (3DAA: paritaprevir/ritonavir - ombitasvir + dasabuvir (ABBVIE REGIMEN) plus RBV) | 140 | 17 | 2 | 0
Completed | 118 | 263 | 40 | 0
Not Completed | 27 | 15 | 8 | 1
Not completed — Did Not Start Treatment | 0 | 0 | 1 | 1
Not completed — Failure to Return | 20 | 10 | 7 | 0
Not completed — Death | 2 | 3 | 0 | 0
Not completed — Other, Not Specified | 5 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: all enrolled participants who received ≥1 dose of ABBVIE REGIMEN, grouped according to treatment regimen (actual treatment received). This presentation was necessary for baseline characteristics since some study-specific measures for which Baseline data are required were analyzed only according to actual treatment received.
Groups:
- 2 DAA+RBV: Two direct-acting antivirals (2DAA): paritaprevir/ritonavir - ombitasvir (ABBVIE REGIMEN) plus RBV
- 3DAA: Three direct-acting antivirals (3DAA): paritaprevir/ritonavir - ombitasvir + dasabuvir (ABBVIE REGIMEN)
- 3DAA+RBV: 3DAA: paritaprevir/ritonavir - ombitasvir + dasabuvir (ABBVIE REGIMEN) plus RBV
- Total: Total of all reporting groups
Arm/Group | 2 DAA+RBV | 3DAA | 3DAA+RBV | Total
Number analyzed (Participants) | 45 | 266 | 159 | 470
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (11.5) | 55 (13.6) | 49 (11.9) | 52 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 124 | 38 | 172
  Male | 35 | 142 | 121 | 298
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 41 | 255 | 152 | 448
  Black | 0 | 2 | 1 | 3
  Asian/Oriental | 4 | 3 | 5 | 12
  Other, Not Specified | 0 | 6 | 1 | 7
Pictorial Representation of Illness and Self-Measure (PRISM) Tool [Mean (Standard Deviation); unit: cm] — PRISM is a visual quantitative method to assess the perceived burden of suffering due to illness. The distance between the center of the "self" (yellow disk) and the illness disk (red disk) is called "self-illness separation" (SIS) and is measured in cm (range is 0 - 27). The smaller the distance, the higher the burden of suffering. Population: participants with a Baseline assessment
  cm
    number analyzed (Participants) | 43 | 263 | 158 | 464
    (all) | 13.1 (9.16) | 12.3 (8.78) | 12.4 (8.89) | 12.4 (8.84)
Chronic Illness Therapy-Fatigue (FACIT-F) Scale [Mean (Standard Deviation); unit: units on a scale] — The FACIT-F Scale is a 13-item questionnaire that assesses self-reported fatigue during the past 7 days and its impact upon daily activities and function. Scores range from 0 - 100, with higher scores indicating a lesser degree of fatigue. Population: participants with a Baseline assessment
  units on a scale
    number analyzed (Participants) | 42 | 256 | 148 | 446
    (all) | 70.8 (22.1) | 69.3 (23.1) | 67.4 (23.1) | 68.8 (23.0)
Patient Activation Measure (PAM-13) Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The PAM-13 item scale is a measure used to assess the patient knowledge, skill, and confidence for self-management. Scores range from 0 to 100. Higher scores indicate and higher level of knowledge, skill and confidence. Population: participants with a Baseline assessment
  units on a scale
    number analyzed (Participants) | 41 | 207 | 139 | 387
    (all) | 64.1 (11.8) | 64.3 (10.1) | 63.0 (9.49) | 63.8 (10.1)
Work Productivity and Activity Impairment (WPAI): Total Work Productivity Impairment [Mean (Standard Deviation); unit: percentage of work productivity impairme] — The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total work productivity impairment indicates the percentage of overall work impairment due to health problems. Population: participants with a Baseline assessment
  percentage of work productivity impairme
    number analyzed (Participants) | 22 | 105 | 58 | 185
    (all) | 14.2 (17.9) | 19.1 (28.0) | 18.1 (23.3) | 18.2 (25.5)
WPAI: Total Activity Impairment [Mean (Standard Deviation); unit: percentage of activity impairment] — The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total activity impairment indicates the percentage of general (non-work) activity impairment due to health problems. Population: participants with a Baseline assessment
  percentage of activity impairment
    number analyzed (Participants) | 43 | 242 | 147 | 432
    (all) | 23.0 (25.8) | 25.9 (27.3) | 28.0 (28.9) | 26.3 (27.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR12)
Description: SVR12 is defined as hepatitis C virus (HCV) ribonucleic acid (RNA) less than the lower limit of quantification (< 50 IU/mL) 12 weeks after the last actual dose of the ABBVIE REGIMEN.
Time Frame: 12 weeks after the last dose of study drug (treatment period was 12 or 24 weeks)
Population: Core Population: Participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype; the prescribed ABBVIE REGIMEN was known) with sufficient follow-up data regarding SVR12.
Measure: Number; unit: percentage of participants
Groups:
- All Participants: Treatment-naïve or -experienced participants with confirmed CHC genotype 1 or 4, receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± RBV according to standard of care and in line with the current local label
- All Genotype 1 Participants: Treatment-naïve or -experienced participants with confirmed CHC genotype 1, receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir with dasabuvir (ABBVIE REGIMEN) ± RBV according to standard of care and in line with the current local label.
- Genotype 1a Participants: Treatment-naïve or -experienced participants with confirmed CHC G1a (includes all GT1-participants except participants with GT1b or GT1b/4), receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir with dasabuvir (ABBVIE REGIMEN) + RBV according to standard of care and in line with the current local label.
Arm/Group | All Participants | All Genotype 1 Participants | Genotype 1a Participants | Genotype 1b Participants | Genotype 4 Participants
Number analyzed (Participants) | 470 | 423 | 145 | 278 | 47
percentage of participants | 88.1 | 88.4 | 77.9 | 93.9 | 85.1

2. Secondary Outcome: Percentage of Participants With Virological Response at End of Treatment (EoTR)
Description: Virological response is defined as HCV RNA < 50 IU/mL. End of Treatment (EoT) is defined as the last intake of ABBVIE REGIMEN or RBV.
Time Frame: EoT, (treatment period was 12 weeks or 24 weeks)
Population: Core Population: Participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype; the prescribed ABBVIE REGIMEN was known).
Measure: Number; unit: percentage of participants
Arm/Group | All Participants | All Genotype 1 Participants | Genotype 1a Participants | Genotype 1b Participants | Genotype 4 Participants
Number analyzed (Participants) | 470 | 423 | 145 | 278 | 47
percentage of participants | 93.4 | 94.8 | 89.0 | 97.8 | 80.9

3. Secondary Outcome: Number of Participants With On-Treatment Virological Failure or Relapse
Description: The number of participants meeting the following SVR12 non-response categories:
  1. On-treatment virological failure (breakthrough) defined >= 1 documented HCV RNA < 50 IU/mL followed by HCV RNA >= 50 IU/mL during treatment or failure to suppress (each measured on-treatment HCV RNA value >= 50 IU/mL)
  2. Relapse defined as HCV RNA < 50 IU/mL at EoT followed by HCV RNA >= 50 IU/mL post-treatment in participants who completed treatment (<= 7 days shortened).
Time Frame: Up to post-treatment Week 12 (treatment period was 12 or 24 weeks)
Population: Core Population: Participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype; the prescribed ABBVIE REGIMEN was known). Participants with non-response 12 weeks after EoT.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants | All Genotype 1 Participants | Genotype 1a Participants | Genotype 1b Participants | Genotype 4 Participants
Number analyzed (Participants) | 56 | 49 | 32 | 17 | 7
Participants
  On-Treatment Virological Failure | 6 | 3 | 3 | 0 | 3
  Relapse | 5 | 5 | 1 | 4 | 0

4. Secondary Outcome: Percentage of Participants With Rapid Virological Response at Week 4 (RVR4)
Description: RVR4 is defined as participants with HCV RNA < 50 IU/mL at Week 4.
Time Frame: Week 4
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | All Participants | All Genotype 1 Participants | Genotype 1a Participants | Genotype 1b Participants | Genotype 4 Participants
Number analyzed (Participants) | 470 | 423 | 145 | 278 | 47
percentage of participants | 57.0 | 57.2 | 62.1 | 54.7 | 55.3

5. Secondary Outcome: Percentage of Participants With Sustained Virological Response 24 Weeks After EoT (SVR24)
Description: SVR24 is defined as HCV RNA < 50 IU/mL 24 Weeks After EoT.
Time Frame: 24 Weeks After EoT (treatment period was 12 or 24 weeks)
Population: Core Population: Participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype; the prescribed ABBVIE REGIMEN was known) with sufficient follow-up data regarding SVR24.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants | All Genotype 1 Participants | Genotype 1a Participants | Genotype 1b Participants | Genotype 4 Participants
Number analyzed (Participants) | 362 | 325 | 97 | 228 | 37
percentage of participants | 95.0 | 95.4 | 92.8 | 96.5 | 91.9

6. Secondary Outcome: Percentage of Participants With Sustained Virological Response 48 Weeks After EoT (SVR48)
Description: SVR48 is defined as participants with HCV RNA < 50 IU/mL 48 weeks after EoT.
Time Frame: 48 Weeks After EoT (treatment period was 12 or 24 weeks)
Population: Core Population: Participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype; the prescribed ABBVIE REGIMEN was known) with sufficient follow-up data regarding SVR48.
Measure: Number; unit: percentage of participants
Groups:
- All Participants: Treatment-naïve or -experienced participants with confirmed chronic hepatitis C (CHC), genotype 1 or 4, receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir with or without dasabuvir (ABBVIE REGIMEN) ± ribavirin (RBV) according to standard of care and in line with the current local label
- Genotype 1 Participants: Treatment-naïve or -experienced participants with confirmed CHC genotype 1, receiving combination therapy with the interferon-free paritaprevir/ritonavir - ombitasvir with dasabuvir (ABBVIE REGIMEN) ± RBV according to standard of care and in line with the current local label.
Arm/Group | All Participants | Genotype 1 Participants | Genotype 1a Participants | Genotype 1b Participants | Genotype 4 Participants
Number analyzed (Participants) | 262 | 237 | 73 | 164 | 25
percentage of participants | 92.7 | 93.2 | 89.0 | 95.1 | 88.0

7. Secondary Outcome: Change From Baseline in PRISM Over Time
Description: PRISM is a visual quantitative method to assess the perceived burden of suffering due to illness. The distance between the center of the "self" (yellow disk) and the illness disk (red disk) is called "self-illness separation" (SIS) and is measured in cm (range is 0 - 27). The smaller the distance, the higher the burden of suffering.
Time Frame: Baseline, 12 and 48 weeks after EoT (treatment period was 12 or 24 weeks)
Population: Core Population: Participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype; the prescribed ABBVIE REGIMEN was known). Participants with a measurement at given time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: cm
Groups:
- 2 DAA+RBV: 2DAA: paritaprevir/ritonavir - ombitasvir (ABBVIE REGIMEN) plus RBV
- 3DAA: 3DAA: paritaprevir/ritonavir - ombitasvir + dasabuvir (ABBVIE REGIMEN)
- 3DAA+RBV: 3DAA: paritaprevir/ritonavir - ombitasvir + dasabuvir (ABBVIE REGIMEN) + RBV
Arm/Group | 2 DAA+RBV | 3DAA | 3DAA+RBV
Number analyzed (Participants) | 30 | 222 | 115
cm
  12 Weeks EoT | 5.41 [2.67 to 8.15] | 7.05 [6.04 to 8.05] | 5.31 [3.91 to 6.71]
  48 Weeks EoT: number analyzed (Participants) | 19 | 135 | 76
  48 Weeks EoT | 10.2 [7.16 to 13.2] | 10.1 [8.93 to 11.2] | 10.3 [8.75 to 11.8]
Statistical Analysis 1: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; Week 12; Test type: Superiority; p = 0.1110, ANCOVA — Between group change comparison: overall. The dependent variable is the change of PRISM from Baseline (Visit-Baseline). The analysis is adjusted for Baseline
Statistical Analysis 2: Comparison: 2 DAA+RBV vs 3DAA; Week 12; Test type: Superiority; p = 0.2704, ANCOVA — Between group change comparison: 3DAA - 2DAA+RBV. The dependent variable is the change of PRISM from Baseline (Visit-Baseline). The analysis is adjusted for Baseline; difference in LS means = 1.64, 95% CI 2-sided [-1.28 to 4.56]
Statistical Analysis 3: Comparison: 2 DAA+RBV vs 3DAA+RBV; Week 12; Test type: Superiority; p = 0.9516, ANCOVA — Between group change comparison: 3DAA+RBV - 2DAA+RBV. The dependent variable is the change of PRISM from Baseline (Visit-Baseline). The analysis is adjusted for Baseline; difference in LS means = -0.09, 95% CI 2-sided [-3.17 to 2.98]
Statistical Analysis 4: Comparison: 3DAA vs 3DAA+RBV; Week 12; Test type: Superiority; p = 0.0489, ANCOVA — Between group change comparison: 3DAA+RBV - 3DAA. The dependent variable is the change of PRISM from Baseline (Visit-Baseline). The analysis is adjusted for Baseline; difference in LS means = -1.73, 95% CI 2-sided [-3.46 to -0.01]
Statistical Analysis 5: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; Week 48; Test type: Superiority; p = 0.9785, ANCOVA — [p-value comment as in outcome 7, analysis 1]
Statistical Analysis 6: Comparison: 2 DAA+RBV vs 3DAA; Week 48; Test type: Superiority; p = 0.9379, ANCOVA — [p-value comment as in outcome 7, analysis 2]; difference in LS means = -0.13, 95% CI 2-sided [-3.37 to 3.11]
Statistical Analysis 7: Comparison: 2 DAA+RBV vs 3DAA+RBV; Week 48; Test type: Superiority; p = 0.9678, ANCOVA — [p-value comment as in outcome 7, analysis 3]; difference in LS means = 0.07, 95% CI 2-sided [-3.33 to 3.47]
Statistical Analysis 8: Comparison: 3DAA vs 3DAA+RBV; Week 48; Test type: Superiority; p = 0.8373, ANCOVA — [p-value comment as in outcome 7, analysis 4]; difference in LS means = 0.20, 95% CI 2-sided [-1.70 to 2.10]
Statistical Analysis 9: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; Week 12 vs Baseline across all participants; Test type: Superiority; p < 0.0001, paired t-test; paired t-test of whether difference in means is 0; Mean Difference (Final Values) = 6.37, 95% CI 2-sided [5.417 to 7.320]
Statistical Analysis 10: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; Week 48 vs Baseline across all participants; Test type: Superiority; p < 0.0001, paired t-test; paired t-test of whether difference in means is 0; Mean Difference (Final Values) = 10.15, 95% CI 2-sided [8.936 to 11.362]

8. Secondary Outcome: Percentage of Participants With ≥ 1 Comorbidity and/or Co-Infection
Time Frame: up to post-treatment Week 48 (treatment period was 12 or 24 weeks)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | All Participants | Genotype 1 Participants | Genotype 1a Participants | Genotype 1b Participants | Genotype 4 Participants
Number analyzed (Participants) | 470 | 423 | 145 | 278 | 47
percentage of participants | 70.0 | 69.3 | 71.0 | 68.3 | 76.6

9. Secondary Outcome: Percentage of Participants Taking ≥ 1 Co-Medication
Time Frame: up to post-treatment Week 48 (treatment period was 12 or 24 weeks)
Population: Safety Population: all enrolled participants who received at least one dose of the ABBVIE REGIMEN (the prescribed ABBVIE REGIMEN was known).
Measure: Number; unit: percentage of participants
Groups:
- Total: * 2DAA: paritaprevir/ritonavir - ombitasvir [ABBVIE REGIMEN]) plus RBV
  * 3DAA: paritaprevir/ritonavir - ombitasvir + dasabuvir [ABBVIE REGIMEN])
  * 3DAA: paritaprevir/ritonavir - ombitasvir + dasabuvir (ABBVIE REGIMEN) plus RBV
Arm/Group | Total | 2 DAA+RBV | 3DAA | 3DAA+RBV
Number analyzed (Participants) | 470 | 45 | 266 | 159
percentage of participants | 59.1 | 64.4 | 54.1 | 66.0

10. Secondary Outcome: Mean Duration of of ABBVIE REGIMEN and RBV Taken
Description: Documented by participant interview and/or participant diary.
Time Frame: Up to Week 12 or Week 24
Population: Safety Population: all enrolled participants who received at least one dose of the ABBVIE REGIMEN (the prescribed ABBVIE REGIMEN was known) and had an assessment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Total | 2 DAA+RBV | 3DAA | 3DAA+RBV
Number analyzed (Participants) | 468 | 45 | 265 | 158
days
  ABBVIE REGIMEN | 83 (11.7) | 84 (3.4) | 83 (9.7) | 84 (15.6)
  RBV: number analyzed (Participants) | 203 | 45 | 0 | 158
  RBV | 81 (18.1) | 84 (3.4) |  | 81 (20.5)

11. Secondary Outcome: Percentage of Planned Duration of ABBVIE REGIMEN and RBV Taken
Description: Planned duration of treatment was 12 or 24 weeks.
Time Frame: Up to Week 12 or Week 24
Population: Core Population: Participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (cirrhotic status, genotype; the prescribed ABBVIE REGIMEN was known). Participants taking specified study drug with non-missing data.
Measure: Mean (Standard Deviation); unit: percentage of planned treatment duration
Arm/Group | All Participants | All Genotype 1 Participants | Genotype 1a Participants | Genotype 1b Participants | Genotype 4 Participants
Number analyzed (Participants) | 468 | 421 | 144 | 277 | 47
percentage of planned treatment duration
  ABBVIE REGIMEN | 98.7 (9.74) | 98.6 (10.18) | 97.7 (12.94) | 99.1 (8.39) | 99.8 (3.91)
  RBV: number analyzed (Participants) | 203 | 156 | 139 | 17 | 47
  RBV | 95.4 (17.55) | 94.1 (19.72) | 95.3 (17.68) | 83.5 (30.68) | 99.8 (3.91)

12. Secondary Outcome: Change From Baseline in FACIT-F Scale Over Time
Description: The FACIT-F Scale is a 13-item questionnaire that assesses self-reported fatigue during the past 7 days and its impact upon daily activities and function. Scores range from 0 - 100, with higher scores indicating a lesser degree of fatigue.
Time Frame: Baseline, EoT (treatment period was 12 or 24 weeks), 12 and 48 weeks after EoT
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 2 DAA+RBV | 3DAA | 3DAA+RBV
Number analyzed (Participants) | 29 | 213 | 112
score on a scale
  EoT | 4.17 [-2.35 to 10.7] | 6.45 [4.05 to 8.86] | 4.49 [1.17 to 7.81]
  12 Weeks EoT: number analyzed (Participants) | 26 | 205 | 107
  12 Weeks EoT | 12.5 [6.78 to 18.3] | 9.92 [7.87 to 12.0] | 10.2 [7.37 to 13.0]
  48 Weeks EoT: number analyzed (Participants) | 13 | 123 | 63
  48 Weeks EoT | 13.3 [4.71 to 22.0] | 9.68 [6.87 to 12.5] | 10.3 [6.37 to 14.3]
Statistical Analysis 1: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; EOT; Test type: Superiority; p = 0.5751, ANCOVA — Between group change comparison: overall. The dependent variable in the change of FACIT-F [0-100] from Baseline (Visit-Baseline). The analysis is adjusted for Baseline
Statistical Analysis 2: Comparison: 2 DAA+RBV vs 3DAA; EoT; Test type: Superiority; p = 0.5176, ANCOVA — Between group change comparison: 3DAA - 2DAA+RBV. The dependent variable in the change of FACIT-F [0-100] from Baseline (Visit-Baseline). The analysis is adjusted for Baseline; difference in LS means = 2.29, 95% CI 2-sided [-4.66 to 9.23]
Statistical Analysis 3: Comparison: 2 DAA+RBV vs 3DAA+RBV; EoT; Test type: Superiority; p = 0.9308, ANCOVA — Between group change comparison: 3DAA+RBV - 2DAA+RBV. The dependent variable in the change of FACIT-F [0-100] from Baseline (Visit-Baseline). The analysis is adjusted for Baseline; difference in LS means = 0.324, 95% CI 2-sided [-7.00 to 7.64]
Statistical Analysis 4: Comparison: 3DAA vs 3DAA+RBV; EoT; Test type: Superiority; p = 0.3462, ANCOVA — Between group change comparison: 3DAA+RBV - 3DAA. The dependent variable in the change of FACIT-F [0-100] from Baseline (Visit-Baseline). The analysis is adjusted for Baseline; difference in LS means = -1.96, 95% CI 2-sided [-6.06 to 2.13]
Statistical Analysis 5: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; 12 Weeks after EoT; Test type: Superiority; p = 0.7016, ANCOVA — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 6: Comparison: 2 DAA+RBV vs 3DAA; 12 weeks after EoT; Test type: Superiority; p = 0.4002, ANCOVA — [p-value comment as in outcome 12, analysis 2]; difference in LS means = -2.61, 95% CI 2-sided [-8.71 to 3.49]
Statistical Analysis 7: Comparison: 2 DAA+RBV vs 3DAA+RBV; 12 weeks after EoT; Test type: Superiority; p = 0.4750, ANCOVA — [p-value comment as in outcome 12, analysis 3]; difference in LS means = -2.33, 95% CI 2-sided [-8.74 to 4.08]
Statistical Analysis 8: Comparison: 3DAA vs 3DAA+RBV; 12 weeks after EoT; Test type: Superiority; p = 0.8740, ANCOVA — [p-value comment as in outcome 12, analysis 4]; difference in LS means = 0.282, 95% CI 2-sided [-3.21 to 3.77]
Statistical Analysis 9: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; 48 weeks after EoT; Test type: Superiority; p = 0.7211, ANCOVA — [p-value comment as in outcome 12, analysis 1]
Statistical Analysis 10: Comparison: 2 DAA+RBV vs 3DAA; 48 weeks after EoT; Test type: Superiority; p = 0.4256, ANCOVA — [p-value comment as in outcome 12, analysis 2]; difference in LS means = -3.67, 95% CI 2-sided [-12.7 to 5.39]
Statistical Analysis 11: Comparison: 2 DAA+RBV vs 3DAA+RBV; 48 weeks after EoT; Test type: Superiority; p = 0.5347, ANCOVA — [p-value comment as in outcome 12, analysis 3]; difference in LS means = -3.01, 95% CI 2-sided [-12.6 to 6.54]
Statistical Analysis 12: Comparison: 3DAA vs 3DAA+RBV; 48 weeks after EoT; Test type: Superiority; p = 0.7920, ANCOVA — [p-value comment as in outcome 12, analysis 4]; difference in LS means = 0.654, 95% CI 2-sided [-4.23 to 5.54]
Statistical Analysis 13: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; Baseline to EOT across all participants; Test type: Superiority; p < 0.0001, paired t-test; paired t-test of mean difference from 0; Mean Difference (Final Values) = 5.64, 95% CI 2-sided [3.355 to 7.935]
Statistical Analysis 14: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; Baseline vs 12 weeks after EOT across all participants; Test type: Superiority; p < 0.0001, paired t-test; paired t-test of mean difference versus 0; Mean Difference (Final Values) = 10.21, 95% CI 2-sided [8.113 to 12.299]
Statistical Analysis 15: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; baseline vs 48 weeks after EOT across all participants; Test type: Superiority; p < 0.0001, paired t-test; paired t-test of mean difference versus 0; Mean Difference (Final Values) = 10.13, 95% CI 2-sided [7.259 to 12.992]

13. Secondary Outcome: Change From Baseline to EoT in PAM-13 Questionnaire
Description: The PAM-13 item scale is a measure used to assess the patient knowledge, skill, and confidence for self-management. Scores range from 0 to 100. Higher scores indicate a higher level of knowledge, skill and confidence.
Time Frame: Baseline, EoT (treatment period was 12 or 24 weeks)
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | 2 DAA+RBV | 3DAA | 3DAA+RBV
Number analyzed (Participants) | 23 | 150 | 93
score on a scale | 1.91 [-1.52 to 5.33] | 0.01 [-1.33 to 1.36] | -0.74 [-2.45 to 0.96]
Statistical Analysis 1: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; Test type: Superiority; p = 0.3869, ANCOVA — Between group change comparison: overall. The dependent variable in the change of PAM-13 from Baseline (Visit-Baseline). The analysis is adjusted for Baseline
Statistical Analysis 2: Comparison: 2 DAA+RBV vs 3DAA; Test type: Superiority; p = 0.3125, ANCOVA — Between group change comparison: 3DAA - 2DAA+RBV. The dependent variable in the change of PAM-13 from Baseline (Visit-Baseline). The analysis is adjusted for Baseline; difference in LS means = -1.89, 95% CI 2-sided [-5.57 to 1.79]
Statistical Analysis 3: Comparison: 2 DAA+RBV vs 3DAA+RBV; Test type: Superiority; p = 0.1741, ANCOVA — Between group change comparison: 3DAA+RBV - 2DAA+RBV. The dependent variable in the change of PAM-13 from Baseline (Visit-Baseline). The analysis is adjusted for Baseline; difference in LS means = -2.65, 95% CI 2-sided [-6.48 to 1.18]
Statistical Analysis 4: Comparison: 3DAA vs 3DAA+RBV; Test type: Superiority; p = 0.4941, ANCOVA — Between group change comparison: 3DAA+RBV - 3DAA. The dependent variable in the change of PAM-13 from Baseline (Visit-Baseline). The analysis is adjusted for Baseline; difference in LS means = -0.76, 95% CI 2-sided [-2.94 to 1.42]
Statistical Analysis 5: Comparison: 2 DAA+RBV vs 3DAA vs 3DAA+RBV; Change from Baseline to Final visit across all participants; Test type: Superiority; p = 0.8842, paired t-test; paired t-test of mean difference vs 0; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-1.271 to 1.096]

14. Secondary Outcome: Change From Baseline Over Time in WPAI: Total Work Productivity Impairment
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total work productivity impairment indicates the percentage of overall work impairment due to health problems.
Time Frame: Baseline, EoT (treatment period was 12 or 24 weeks),12 and 24 weeks after EoT
Population: Core Population: Participants who were adequately treated according to the standard of care and within local label recommendations for their specific disease characteristics (the prescribed ABBVIE REGIMEN was known). Overall: participants with a measurement at Baseline; data rows = participants with a measurement at Baseline and given time point.
Measure: Mean (Standard Deviation); unit: percentage of overall work impairment
Groups:
- Total: 2DAA: paritaprevir/ritonavir - ombitasvir (ABBVIE REGIMEN) plus RBV or 3DAA: paritaprevir/ritonavir - ombitasvir + dasabuvir [ABBVIE REGIMEN]) or 3DAA: paritaprevir/ritonavir - ombitasvir + dasabuvir (ABBVIE REGIMEN) + RBV
Arm/Group | Total | 2 DAA+RBV | 3DAA | 3DAA+RBV
Number analyzed (Participants) | 185 | 22 | 105 | 58
percentage of overall work impairment
  EoT: number analyzed (Participants) | 126 | 16 | 68 | 42
  EoT | 5.5 (31.4) | 5.0 (36.4) | 4.4 (27.1) | 7.5 (36.3)
  12 Weeks EoT: number analyzed (Participants) | 113 | 11 | 68 | 34
  12 Weeks EoT | -4.3 (23.4) | -4.2 (11.9) | -3.8 (21.5) | -5.4 (29.6)
  24 Weeks EoT: number analyzed (Participants) | 99 | 11 | 63 | 25
  24 Weeks EoT | -7.4 (22.1) | -3.2 (33.6) | -7.2 (22.1) | -9.7 (15.6)

15. Secondary Outcome: Change From Baseline Over Time in WPAI: Total Activity Impairment
Description: The WPAI Hepatitis C V2.0 is an HCV specific questionnaire used to measure work absenteeism, work presenteeism, and daily activity impairment. Respondents were asked about time missed from work and time while at work during which productivity was impaired in the past seven days. Results of WPAI are expressed as a percentage of impairment from 0 to 100, with higher percentages indicating greater impairment and less productivity.
  Total activity impairment indicates the percentage of general (non-work) activity impairment due to health problems.
Time Frame: Baseline, EoT (treatment period was 12 or 24 weeks),12 and 24 weeks after EoT
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: percentage impairment of activity
Arm/Group | Total | 2 DAA+RBV | 3DAA | 3DAA+RBV
Number analyzed (Participants) | 432 | 43 | 242 | 147
percentage impairment of activity
  EoT: number analyzed (Participants) | 322 | 27 | 194 | 101
  EoT | -2.1 (30.9) | 7.0 (25.2) | -3.0 (28.9) | -2.8 (35.5)
  12 Weeks EoT: number analyzed (Participants) | 317 | 26 | 189 | 102
  12 Weeks EoT | -11.9 (27.0) | -7.7 (22.0) | -13.3 (24.8) | -10.5 (31.6)
  24 Weeks EoT: number analyzed (Participants) | 275 | 23 | 170 | 82
  24 Weeks EoT | -13.4 (25.9) | -11.3 (22.8) | -12.3 (24.0) | -16.3 (30.3)

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs and/or Pregnancies
Description: An adverse event (AE) is defined as any untoward medical occurrence. If an AE meets any of the following criteria, it is considered serious: results in death, is life threatening, results in hospitalization or prolongation of hospitalization, is a congenital anomaly, results in significant disability/incapacity, or is an important medical event. TEAEs are defined as any reported event that begins or worsens in severity after initiation of study drug through 30 days post-study drug dosing.
Time Frame: up to 30 days post treatment (treatment period was 12 weeks or 24 weeks)
Population: Safety Population: all enrolled participants who received at least one dose of the ABBVIE REGIMEN (the prescribed ABBVIE REGIMEN was known). Pregnancy data presented for female participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | Total | 2 DAA+RBV | 3DAA | 3DAA+RBV
Number analyzed (Participants) | 470 | 45 | 266 | 159
Participants
  ≥ 1 TEAE | 124 | 16 | 65 | 43
  ≥ 1 Serious TEAE | 13 | 1 | 7 | 5
  Pregnancy: number analyzed (Participants) | 172 | 10 | 124 | 38
  Pregnancy | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 30 days post treatment (treatment period was 12 weeks or 24 weeks)
Description: Treatment-emergent AEs are presented. Treatment-emergent AEs are defined as any reported AE that begins or worsens in severity after initiation of study drug through 30 days after last study drug intake.
  Treatment duration was not a factor for assignment to reporting groups.
Arm/Group | 2 DAA+RBV | 3DAA | 3DAA+RBV
All-Cause Mortality (participants affected / at risk) | 0/45 | 4/266 | 1/159
Serious Adverse Events (participants affected / at risk) | 1/45 | 7/266 | 5/159
Other Adverse Events (participants affected / at risk) | 7/45 | 33/266 | 23/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 DAA+RBV (N=45) | 3DAA (N=266) | 3DAA+RBV (N=159)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
GASTRIC PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
HEPATIC CIRRHOSIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
OROPHARYNGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
BLOOD POTASSIUM DECREASED (Investigations) | 0 (0) | 1 (1) | 0 (0)
PSEUDARTHROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2 DAA+RBV (N=45) | 3DAA (N=266) | 3DAA+RBV (N=159)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 8 (8)
FATIGUE (General disorders) | 2 (2) | 21 (21) | 9 (9)
HEADACHE (Nervous system disorders) | 0 (0) | 15 (15) | 4 (4)
RASH (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/45/NCT02615145/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT02615145/SAP_001.pdf